CLINICAL TRIAL: NCT07067255
Title: Phase 1/2 Study of Sequential CD146 and GPC3 CAR-T Cell Therapy in Advanced Ovarian Cancer
Brief Title: Sequential CD146 and GPC3 CAR-T Cell Therapy in Advanced Ovarian Cancer
Acronym: BAH2573-104
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Essen Biotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESBI202571-104
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Cancer; Ovarian Carcinoma; Ovarian Sarcoma; Ovarian Cancer Stage IV
Keywords: GPC3; CD146; CRISPR-Cas9; CAR-T; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients enrolled in this clinical trial will receive a carefully designed treatment regimen. Before the infusion of CD146 and GPC3 CAR-T cells, participants will undergo preconditioning chemotherapy. This chemotherapy serves to create an optimal environment for CAR-T cell therapy to effectively target and eliminate cancer cells. Following chemotherapy, participants will receive the infusion of CD146 and GPC3 CAR-T cells.
Masking Description: Open-label clinical trials are a category of clinical research where the masking is minimal or nonexistent. In such trials, both the participants and the researchers are fully aware of the treatment assignments, which means participants know the treatment they are receiving, and researchers are aware of each participant's treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD146 GPC3 CAR T cells, chemotherapy (Experimental): Patients will be administered fludarabine phosphate intravenously (IV) over a 30-minute period on days -4 to -2. Additionally, cyclophosphamide will be administered intravenously (IV) over 60 minutes on day -2. Subsequently, patients will receive CD146 GPC3 CAR T cells intravenously (IV) over a duration of 10-20 minutes on day 0. Patients who exhibit positive responses to the initial dose of GPC3 /CD146 CAR T cells, do not experience unacceptable side effects, and have a sufficient quantity of cells available may be eligible to receive 2 or 3 additional doses of GPC3/CD146 CAR T cells.
  Interventions: Biological: GPC3 CD146 CAR-T cells

INTERVENTIONS:
Biological: GPC3 CD146 CAR-T cells — The intervention in this clinical trial involves a novel approach using CD146/GPC3 Chimeric Antigen Receptor T (CAR T) cells combined with chemotherapy. The goal is to assess safety and efficacy in patients with specific hematologic malignancies.
  Treatment Regimen:
  Patients in the trial will undergo the following regimen:
  Fludarabine Phosphate (Days -4 to -2): IV administration of fludarabine phosphate over 30 minutes on days -4 to -2. It's part of the preparatory regimen to enhance the body's response to CAR T-cell therapy.
  Cyclophosphamide (Day -2): IV cyclophosphamide over 60 minutes on day -2.
  GPC3/CD146 Chimeric Antigen Receptor T Cells (Day 0): IV administration of investigational therapy, GPC3/CD146 CAR T cells, over 10-20 minutes on day 0.
  Additional Doses: Eligible patients responding well to the initial CD146/GPC3 CAR-T cell infusion without unacceptable side effects and sufficient CAR-T cell availability may receive 2 or 3 additional doses.

SUMMARY:
This is a multicenter, open-label Phase 1/2 clinical trial evaluating the safety and preliminary efficacy of sequentially administered CD146-targeted and GPC3-targeted CAR-T cell therapy in patients with advanced relapsed or refractory ovarian cancer. Eligible patients will undergo lymphodepleting chemotherapy with cyclophosphamide and fludarabine, followed by an infusion of autologous CD146-directed CAR-T cells (Arm A) and a subsequent infusion of autologous GPC3-directed CAR-T cells (Arm B). The Phase 1 portion will assess safety, tolerability, and dose-limiting toxicities (DLTs) to determine a recommended Phase 2 dose, while the Phase 2 portion will evaluate efficacy endpoints including objective response rate (ORR), progression-free survival (PFS), and overall survival (OS). Patients will be followed for up to 36 months after CAR-T infusion to monitor long-term outcomes and adverse events.

DETAILED DESCRIPTION:
Advanced ovarian cancer remains challenging to treat, especially in the relapsed or refractory setting. CD146 (also known as MUC18 or MCAM) is a cell adhesion molecule involved in tumor angiogenesis and metastasis; it is frequently overexpressed in ovarian cancer and has been associated with aggressive disease and poor prognosis. GPC3 (glypican-3) is an oncofetal antigen expressed in a subset of ovarian carcinomas (particularly clear cell histology) and has been identified as a potential immunotherapy target in ovarian cancer. By targeting both CD146 and GPC3, this dual CAR-T approach aims to address tumor heterogeneity and improve anti-tumor efficacy. Essen Biotech's CAR-T pipeline emphasizes multi-target strategies (including CD146) and innovative dual-CAR designs to overcome the solid tumor microenvironment, providing the rationale for sequentially administering two distinct CAR-T cell products in this study.

In the Phase 1 portion (dose escalation), patients will be enrolled in sequential cohorts to receive escalating doses of CD146 CAR-T cells followed by GPC3 CAR-T cells. A standard 3+3 dose escalation design may be used to identify the maximum tolerated dose (MTD) and any dose-limiting toxicities. Lymphodepleting conditioning with cyclophosphamide and fludarabine will be given prior to CAR-T infusion to enhance T-cell engraftment. Arm A consists of an infusion of CD146-targeted CAR-T cells at the assigned dose; after a short interval (e.g. 1-7 days), Arm B consists of an infusion of GPC3-targeted CAR-T cells. Patients are closely monitored during and after each infusion for acute toxicities, including cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS). The DLT observation period is typically the first 28 days following the sequential CAR-T infusions. If DLTs occur, dose levels may be adjusted accordingly. Once the Phase 1 portion establishes a recommended Phase 2 dose, the trial will expand into the Phase 2 portion.

In the Phase 2 expansion, additional patients will be treated at the established dose to further evaluate efficacy outcomes. Tumor response will be assessed by imaging (e.g. RECIST 1.1 criteria) at regular intervals. The primary endpoints in Phase 2 include Objective Response Rate (the proportion of patients achieving a complete or partial response). Secondary efficacy endpoints include Progression-Free Survival (time from CAR-T infusion to disease progression or death) and Overall Survival (time from CAR-T infusion to death from any cause). Patients will also be evaluated for duration of response and immunological correlative endpoints (such as CAR-T cell persistence in blood), as applicable. All participants will be followed for up to 36 months post-treatment for long-term safety surveillance and survival status. This trial design will provide critical initial data on the feasibility, safety profile, and potential anti-tumor activity of a sequential dual-CAR T-cell therapy in ovarian cancer patients who have exhausted standard therapies.

ELIGIBILITY:
Inclusion Criteria:

* Expected survival time ≥3 months;
* Diagnosis: Histologically or cytologically confirmed epithelial ovarian carcinoma (including fallopian tube or primary peritoneal carcinoma considered as ovarian cancer) that is relapsed or refractory to standard therapies. Patients must have received and progressed on or after at least one line of platinum-based chemotherapy (or be platinum-resistant) and have no curative standard treatment options.
* Target Antigen Expression: Tumor must demonstrate positive expression of CD146 and GPC3 by immunohistochemistry (IHC) on a recent tumor tissue sample. Expression of both targets is required for eligibility (to ensure the presence of the CAR-T targets in the patient's cancer).
* Disease Status: Measurable disease as defined by RECIST 1.1 criteria (at least one measurable lesion on imaging).
* Age: Adults aged ≥18 years. (Patients must be legally adult and able to provide informed consent. Upper age limit may not be specified, but patients must meet other health criteria.)
* Performance Status: Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (indicative of fully active or restricted in physically strenuous activity only).
* Organ Function: Adequate organ and bone marrow function, including: absolute neutrophil count (ANC) above a minimum threshold, platelet count above threshold, hemoglobin above threshold (transfusion allowed), serum AST/ALT and bilirubin ≤2× upper limit of normal (unless due to liver involvement by tumor), and adequate renal function (e.g. creatinine clearance ≥50 mL/min or per protocol criteria).
* Consent: Ability to understand and sign informed consent, and willing to comply with trial procedures and follow-up. Women of child-bearing potential must have a negative pregnancy test and agree to use effective contraception during the study and for a defined period after CAR-T cell infusion (due to unknown risks to a fetus).

Exclusion Criteria:

* Prior Therapy: Previous treatment with any CAR-T cell therapy or other gene-engineered T-cell therapy targeting CD146 or GPC3. (Patients who received prior immunotherapies such as checkpoint inhibitors are allowed if a washout period is met, but prior CAR-T could confound results or pose increased risk.)
* CNS Involvement: Active central nervous system (CNS) metastases or carcinomatous meningitis. (Patients with a history of CNS metastases that have been effectively treated and are radiographically stable off steroids may be eligible, per protocol specifics.)
* Comorbid Illness: Uncontrolled intercurrent illness including, but not limited to, active uncontrolled infection, clinically significant heart failure (e.g. NYHA Class III-IV), unstable angina or arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. (Patients with controlled chronic conditions may be eligible at the investigator's discretion.)
* Immunosuppression: Active hepatitis B or C infection with viremia, or known HIV infection with uncontrolled viral load. Patients requiring chronic systemic immunosuppressive therapy (e.g. for an autoimmune condition or organ transplant) are excluded, except for physiologic dose steroids.
* Pregnancy or Breastfeeding: Pregnant or breastfeeding women are excluded due to potential risks to the fetus or infant from the study treatment. Women of child-bearing potential who are unwilling or unable to use adequate contraception are not eligible.
* Other Malignancy: Presence of another active malignancy requiring treatment (with the exception of certain early-stage cancers or those in remission for a specified period, per protocol). This is to avoid confounding outcomes and ensure patient safety.
* Hypersensitivity: Known severe hypersensitivity to any component of the investigational CAR-T cell products or to the lymphodepletion chemotherapy drugs (cyclophosphamide, fludarabine).
* Other Exclusions: Any condition that, in the opinion of the investigator, would make the patient unsuitable for the study (such as life expectancy limited by comorbid illness, or significant laboratory abnormalities not covered above).

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2028-12-10 (Estimated); Study Completion 2029-12-28 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose-limiting toxicities (DLTs) following chemotherapy preparative regimen and infusion of GPC3/CD146 chimeric antigen receptor (CAR) T cells | 28 days
  Will be recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 at three dose levels until the maximum tolerated dose (MTD) is determined.

SECONDARY OUTCOMES:
Rate of successful manufacture and expansion of the CD146/GPC3 chimeric antigen receptor (CAR) T cells | 60 days
  satisfy the targeted dose level and meet the required release specifications outlined in the Certificate of Analysis (COA)

CONTACTS AND LOCATIONS:
Locations (1):
- District One Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No